CLINICAL TRIAL: NCT01312818
Title: A Therapeutic Trial of Bortezomib (Velcade), Vorinostat (SAHA) and Dexamethasone for Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL)
Brief Title: Bortezomib, Vorinostat and Dexamethasone for Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008LS113; MT2008-33R (Other: Blood and Bone Marrow Transplantation Program); 1010M91973 (Other: IRB, University of Minnesota); X05323 (Other: Millennium Pharmaceuticals, Inc.)
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib; Vorinostat; Dexamethasone; Calcium Dobesilate; Methotrexate; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): Bortezomib IV Vorinostat PO Dexamethasone PO Intrathecal Methotrexate Imatinib Mesylate PO (for Ph+ ALL patients only)
  Interventions: Drug: Bortezomib; Drug: Vorinostat; Drug: Dexamethasone; Drug: Methotrexate; Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Bortezomib — 1.3 mg/m^2 by intravenous pyelogram (IVP) over 3-5 seconds on days 1, 4, 8 and 11.
  Other Names: Velcade(R)
Drug: Vorinostat — 180 mg/m^2 (max dose 400mg) by mouth (PO) divided twice a day (BID) on days 1-14
  Other Names: suberoylanilide hydroxamic acid (SAHA); Zolinza
Drug: Dexamethasone — 6 mg/m^2 by mouth (PO) divided twice a day (BID) on days 4-15.
  Other Names: Decadron
Drug: Methotrexate — Intrathecal Methotrexate at age based dose on day 1 (repeat on day 15 or 16 for CNS positive patients only)
  Other Names: Trexall; amethopterin
Drug: Imatinib mesylate — For Ph+ acute lymphoblastic leukemia (ALL) patients only:
  Imatinib Mesylate is allowable at 340 mg/m2 PO once a day (rounded to the nearest 100 mg) for age ≤18 years and 400 mg for >18 years on Days 1-16.
  Other Names: Gleevec(R)

SUMMARY:
Both of bortezomib and vorinostat have identified Phase II doses for pediatric and adult patients of which no grade 4 dose limiting toxicities have been observed in prior studies. The pre-clinical synergy of these 2 agents when used in combination along with the lack of over-riding toxicities and different mechanisms of action provide strong rationale for a clinical trial investigating bortezomib and vorinostat in combination. This trial will use the identified Phase II dose which is at or below the maximum tolerated dose for both agents which have very acceptable toxicity profiles and such should prove feasible and tolerable in this relapsed/refractory ALL population.

DETAILED DESCRIPTION:
This is a phase II study of bortezomib 1.3 mg/m^2 by intravenous pyelogram (IVP) on days 1, 4, 8, and 11, vorinostat 180 mg/m^2 by mouth (PO) per day (not to exceed 400 mg per day) days 1-14, and dexamethasone 6 mg/m^2 PO days 4-15 for the treatment of relapsed/refractory acute lymphoblastic leukemia (ALL). No more than 3 treatment courses may be given.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of lymphoblastic lymphoma or acute lymphoblastic leukemia (ALL) with ≥ 5% blasts in the bone marrow (M2/M3) with or without extramedullary disease that meets one of the following criteria:

  * Refractory Disease/Induction Failure: Failure to achieve initial remission after 2 attempts of standard induction therapy
  * Relapsed Disease: Patients in relapse #1 or higher for whom standard curative therapies or therapies to prolong survival do not exist.

Patients who are Philadelphia chromosome-positive (Ph + ALL) are eligible provided they are not imatinib resistant or intolerant.

Patients with CNS positive disease will be eligible.

* Age 2 to 30 years
* Karnofsky ≥ 50% for patients 16 years and older and Lansky status ≥ 50 for patients under 16 years of age.
* Patients must have a life expectancy ≥ 8 weeks as determined by the enrolling investigator.
* Have acceptable organ function as defined within 7 days of starting treatment:

  * Renal: creatinine clearance ≥ 70ml/min/1.73m^2 or serum creatinine based on age/gender as follows: Maximum serum creatinine (mg/dl) 0.8 for 2 years to <6 years; 1.0 for 6 years to <10 years; 1.2 for 10 years to <13 years; 1.5 male and 1.4 female for 13 years to <16 years; 1.7 male and 1.4 female for ≥ 16 years
  * Hepatic: ALT < 5 x upper limit of normal (ULN) and total bilirubin ≤ 1.5x upper limit of normal (ULN) for age.
  * Cardiac: left ventricular ejection fraction ≥ 40% by echocardiogram/multi gated acquisition scan (ECHO/MUGA). Normal QTc on electrocardiogram (EKG) (not to exceed upper limit of normal - men: 430 milliseconds (ms); women: 450 ms; children up to 15 years: 440 ms).
* Prior Therapy:

  * Patients must have recovered from the non-hematologic toxic effects of all prior therapy before entry onto this trial. Recovery is defined as a Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 toxicity grade <2, unless otherwise specified in the Inclusion and Exclusion Criteria.

Cytotoxic therapy: Patients must have had their last dose of chemotherapy at least two weeks prior to study entry.

* Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor and at least 14 days since pegfilgrastim (Neulasta®) administration.
* Biologic (anti-neoplastic) therapy: At least 7 days since the completion of therapy with a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair.
* Monoclonal antibodies: At least 3 half-lives of the antibody after the last administration of a monoclonal antibody.
* Hematopoietic Stem Cell Transplant (HSCT): Patients who have experienced their relapse after a HSCT are eligible, provided they have no evidence of Graft-versus-Host Disease (GVHD).

  * Women of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment and for 2 months after the last dose of chemotherapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment and for 2 months after the last dose of chemotherapy.
  * Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject/guardian at any time without prejudice to future medical care.

Exclusion Criteria:

* Pregnant or lactating. The agents used in this study are known to be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for surgically sterilized women.
* Known hypersensitivity to bortezomib, boron or mannitol or any of the agents or their ingredients used in this study.
* Inability to swallow capsules.
* Grade 2 or greater peripheral neuropathy within 14 days before study registration.
* Patients with untreated positive blood cultures or progressive infections as assessed by radiographic studies.
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (appendix VI), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Serious concomitant medical or psychiatric disorders (e.g., active infection, uncontrolled diabetes) that, in the opinion of the investigator, would compromise the safety of the patient or likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Patient has received investigational drugs within the 14 days before study registration.
* Radiation therapy within 3 weeks before registration. Enrollment of patients who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Burke, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University if Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy: bortezomib, vorinostat and dexamethasone combination, as well as intrathecal methotrexate and imatinib mesylate.
  Bortezomib: 1.3 mg/m^2 by intravenous pyelogram (IVP) over 3-5 seconds on days 1, 4, 8 and 11.
  Vorinostat: 180 mg/m^2 (max dose 400mg) by mouth (PO) divided twice a day (BID) on days 1-14
  Dexamethasone: 6 mg/m^2 by mouth (PO) divided twice a day (BID) on days 4-15.
  Methotrexate: Intrathecal Methotrexate at age based dose on day 1 (repeat on day 15 or 16 for CNS positive patients only)
  Imatinib mesylate: For Ph+ acute lymphoblastic leukemia (ALL) patients only:
  Imatinib Mesylate is allowable at 340 mg/m2 PO once a day (rounded to the nearest 100 mg) for age ≤18 years and 400 mg for >18 years on Days 1-16.
Period: Overall Study
Arm/Group | Chemotherapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved Complete Remission of Their Disease
Description: Complete Remission (CR): A CR requires that the following be recorded concurrently: an absolute neutrophil count (segs and bands) > 1000/μL, no circulating blasts, platelets > 100,000/μL; adequate bone marrow cellularity with trilineage hematopoiesis, and < 5% marrow leukemia blast cells. All previous extramedullary manifestations of disease must be absent. If patients continue on with treatment, there can be no evidence of recurrence of ALL for at least 4 weeks.
Time Frame: Day 30
Measure: Number; unit: participants
Groups:
- ALL Treated Patients: bortezomib, vorinostat and dexamethasone combination, as well as intrathecal methotrexate and imatinib mesylate.
  Bortezomib: 1.3 mg/m^2 by intravenous pyelogram (IVP) over 3-5 seconds on days 1, 4, 8 and 11.
  Vorinostat: 180 mg/m^2 (max dose 400mg) by mouth (PO) divided twice a day (BID) on days 1-14
  Dexamethasone: 6 mg/m^2 by mouth (PO) divided twice a day (BID) on days 4-15.
  Methotrexate: Intrathecal Methotrexate at age based dose on day 1 (repeat on day 15 or 16 for CNS positive patients only)
  Imatinib mesylate: For Ph+ acute lymphoblastic leukemia (ALL) patients only:
  Imatinib Mesylate is allowable at 340 mg/m2 PO once a day (rounded to the nearest 100 mg) for age ≤18 years and 400 mg for >18 years on Days 1-16.
Arm/Group | ALL Treated Patients
Number analyzed (Participants) | 2
participants | 0

2. Secondary Outcome: Number of Subjects Experiencing Drug Related Adverse Events
Description: To characterize the toxicities of bortezomib, vorinostat and dexamethasone when used in combination. Toxicity will be graded using the NCI's Common Terminology Criteria for Adverse Events (CTCAE 4.0).
Time Frame: Day 1 of Treatment to 30 Days Post Treatment
Measure: Number; unit: participants
Groups:
- ALL Treated Patients: List of toxicities in acute lymphoblastic leukemia (ALL) patients treated with bortezomib, vorinostat and dexamethasone combination, as well as intrathecal methotrexate and imatinib mesylate.
  Bortezomib: 1.3 mg/m^2 by intravenous pyelogram (IVP) over 3-5 seconds on days 1, 4, 8 and 11.
  Vorinostat: 180 mg/m^2 (max dose 400mg) by mouth (PO) divided twice a day (BID) on days 1-14
  Dexamethasone: 6 mg/m^2 by mouth (PO) divided twice a day (BID) on days 4-15.
  Methotrexate: Intrathecal Methotrexate at age based dose on day 1 (repeat on day 15 or 16 for CNS positive patients only)
  Imatinib mesylate: For Ph+ acute lymphoblastic leukemia (ALL) patients only:
  Imatinib Mesylate is allowable at 340 mg/m2 PO once a day (rounded to the nearest 100 mg) for age ≤18 years and 400 mg for >18 years on Days 1-16.
Arm/Group | ALL Treated Patients
Number analyzed (Participants) | 2
participants | 1

3. Secondary Outcome: Number of Subjects With Activated Caspases and Other Regulators of Apoptosis
Description: Activation of caspases and other regulators of apoptosis in treated blast cells will be determined by Western analysis (correlative lab analysis).
Time Frame: From Day 1 to 30 Days After Last Dose
Population: The trial was terminated early with only 2 patients so caspase samples were not sent for analysis.
Groups:
- Chemotherapy: Bortezomib IV Vorinostat PO Dexamethasone PO Intrathecal Methotrexate Imatinib Mesylate PO (for Ph+ ALL patients only)
  Bortezomib: 1.3 mg/m^2 by intravenous pyelogram (IVP) over 3-5 seconds on days 1, 4, 8 and 11.
  Vorinostat: 180 mg/m^2 (max dose 400mg) by mouth (PO) divided twice a day (BID) on days 1-14
  Dexamethasone: 6 mg/m^2 by mouth (PO) divided twice a day (BID) on days 4-15.
  Methotrexate: Intrathecal Methotrexate at age based dose on day 1 (repeat on day 15 or 16 for CNS positive patients only)
  Imatinib mesylate: For Ph+ acute lymphoblastic leukemia (ALL) patients only:
  Imatinib Mesylate is allowable at 340 mg/m2 PO once a day (rounded to the nearest 100 mg) for age ≤18 years and 400 mg for >18 years on Days 1-16.
Arm/Group | Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=2)
Sepsis (Infections and infestations) | 1 (1)
death from disease (Blood and lymphatic system disorders) | 1 (1)
esophageal ulcer (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Investigations - Other, specify: hyperphosphatemia (Investigations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No